CLINICAL TRIAL: NCT00862706
Title: An Open-label, Single-arm, Multicenter, Study of Telbivudine in Nucleos(t)Ide-naïve Subjects of Black/African American or Hispanic/Latino Origin With Compensated Chronic Hepatitis B Virus (HBV) Infection
Brief Title: Efficacy of Telbivudine in Blacks/African Americans and Hispanics/Latinos With Compensated Chronic Hepatitis B During 52 Weeks
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Stopped with Patients
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDT600AUS06
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Compensated Chronic Hepatitis B
Keywords: Chronic HBV
MeSH Terms: interventions — Telbivudine

ARMS (1):
- A (Experimental)
  Interventions: Drug: Telbivudine/LDT600A

INTERVENTIONS:
Drug: Telbivudine/LDT600A — Oral once daily

SUMMARY:
The purpose of this study is to investigate the efficacy of telbivudine in Blacks/African Americans and Hispanics/Latinos with compensated chronic hepatitis B during 52 weeks of treatment

ELIGIBILITY:
Inclusion criteria:

1. Patients must give written informed consent before any assessment is performed.
2. Male or female, 16 to 70 years of age.
3. Black/African American race and/or Hispanic/Latino ethnicity
4. Documented compensated chronic hepatitis B defined by all of the following:

   * Clinical history compatible with compensated chronic hepatitis B.
   * Positive serum HBsAg at least 6 months prior to study entry
   * HBeAg-positive or HBeAg-negative at the Screening visit.
   * Detectable serum HBsAg at the Screening visit.
   * Serum ALT level > or = 1.3 and <10x ULN at the Screening visit.
5. Serum HBV DNA level > or = 5 log10 copies/mL as determined by the COBAS™ Amplicor HBV PCR assay at the central study laboratory
6. Willing and able to comply with the study drug regimen and all other study requirements.

Exclusion criteria:

1. Subject is pregnant or breastfeeding. Women of childbearing potential must have a negative serum beta-human chorionic gonadotropin (β-HCG) at Screening.
2. Subject is of reproductive potential (men and women) and unwilling to use double barrier method of contraception. It is required that double barrier method of contraception be used (i.e. condom with spermicide or diaphragm with spermicide) by subjects of reproductive potential (men and women) regardless of whether a hormonal agent is also used as a method of contraception.
3. Subject is co-infected with hepatitis C virus (HCV), hepatitis D virus (HDV), or human immunodeficiency virus (HIV-1 or HIV-2). Patients will be tested for antibodies to HCV, HDV, and HIV at the Screening visit in assessments performed at the central laboratory.
4. Subject previously received lamivudine, adefovir dipivoxil, entecavir, telbivudine or an investigational anti-HBV nucleoside or nucleotide analog at any time. Precluded therapies include, but are not limited to, the following: any previous exposure to lamivudine, adefovir or other PMEA analogs (tenofovir, MCC-478), lobucavir, entecavir, emtricitabine (FTC), L-FMAU, L-Fd4C, or other investigational anti-HBV nucleosides/nucleotides.
5. Subject has received interferon or other immunomodulatory treatment for HBV infection in the 12 months before Screening for this study. Precluded therapies include, but are not limited to, interferon agents (alpha-, beta- or gamma-interferons), thymosin, IL-12, or other putative systemic immunomodulators.
6. Subject has a history of or clinical signs/symptoms of hepatic decompensation such as ascites, variceal bleeding, hepatic encephalopathy, or spontaneous bacterial peritonitis.
7. Subject has a medical condition that requires prolonged or frequent use of systemic acyclovir or famciclovir (e.g., for recurrent herpes virus infections, etc). Prolonged use means episodic treatment with these agents for periods exceeding 10 days every 3 months, or chronic suppressive therapy.
8. Subject has a history of hepatocellular carcinoma (HCC) or findings suggestive of possible HCC, such as suspicious foci on imaging studies or elevated serum alpha-fetoprotein (AFP) levels. In patients with such findings, HCC must be ruled-out prior to Screening for the present study.
9. Subject has one or more additional known primary or secondary causes of liver disease, other than hepatitis B (e.g., alcoholism, autoimmune hepatitis, malignancy with hepatic involvement, hemochromatosis, alpha-1 antitrypsin deficiency, Wilson's Disease, other congenital or metabolic conditions affecting the liver, congestive heart failure or other severe cardiopulmonary disease, etc.). Gilbert's syndrome and Dubin-Johnson syndrome, two benign disorders associated with low-grade hyberbilirubinemia, will not exclude patients from participation in this trial.
10. Subject has a history of clinical or laboratory evidence of pancreatitis or demonstrates a clinical or laboratory course consistent with pancreatitis within 12 weeks of study screening.
11. Subject is currently abusing alcohol or illicit drugs, or has a history of alcohol abuse or illicit substance abuse within the preceding two years. For the purposes of the present study, alcohol abuse is arbitrarily defined as frequent consumption of alcoholic beverages with an average daily intake of more than 40g of ethanol or 3 beers or the equivalent. Patients currently on methadone maintenance treatment programs are NOT eligible for this study due to potential interference with the study evaluations.
12. Subject has a medical condition that requires frequent or prolonged use of systemic corticosteroids (e.g., severe asthma, severe arthritis or autoimmune conditions, organ transplantation, adrenal insufficiency, etc).
13. Subject has any other concurrent medical or social condition likely to preclude compliance with the schedule of evaluations in the protocol, or likely to confound the efficacy or safety observations of the study (e.g., concurrent malignancy; history of unstable angina or repeated myocardial infarction; uncontrolled asthma or diabetes; unstable thyroid disease or other significant hormonal condition; frequent or uncontrolled seizure disorder; severe psychiatric disorder requiring psychotropic medication; active tuberculosis, pneumonia, or other severe infection under current treatment; lives in a country other than that of the investigative site; or has other medical or social circumstances likely to interfere with the schedule of evaluations).
14. A history of treated malignancy (other than hepatocellular carcinoma) is allowable if the subject's malignancy has been in complete remission, off chemotherapy and without additional surgical intervention, during the preceding 3 years.
15. Subject has a history of myopathy, myositis, or persistent muscle weakness or peripheral neuropathy (polyneuropathy).
16. Subject has a known history of allergy to nucleoside analogues.
17. Subject is enrolled or plans to enroll in another clinical trial of an investigational agent while participating in this study.
18. Subject has any of the following laboratory values at Screening:

    * Absolute neutrophil count (ANC) <1500/mm3
    * Hemoglobin <11.0 g/dL (men) or <10.0 g/dL (women)
    * Platelet count <75,000/mm3
    * ALT (SGPT) >10x ULN
    * Serum creatinine >1.5x ULN
    * Total bilirubin >2.0x mg/dL
    * Prothrombin time >2.0 seconds above ULN
    * Serum amylase or lipase > or = 1.5x ULN
    * Serum albumin <3.3 g/dL
    * Serum alpha-fetoprotein (AFP) >50 ng/mL. If AFP is >50 ng/mL, the subject must have an imaging study of the liver demonstrating no evidence of tumor within 60 days prior to study entry.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
non detectable HBV DNA level | week 52

SECONDARY OUTCOMES:
Mean and median reduction in HBV DNA | weeks 2, 4, 8, 12, 16, 24, 32, 40, 48 and 52 or premature D/C
Mean and median reduction from Baseline in absolute ALT level | weeks 2, 4, 8, 12, 16, 24, 32, 40, 48 and 52 or premature D/C
Proportion of patients with ALT normalization | weeks 2, 4, 8, 12, 16, 24, 32, 40, 48 and 52 or premature D/C
Proportion of patients with non-detectable serum HBV DNA | week 24
of patients with HBeAg loss in subjects who were HBeAg positive at Baseline | Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48 and 52 or premature D/C
Proportion of patients with HBeAg seroconversion in subjects who were HBeAg positive at Baseline | 2, 4, 8, 12, 16, 24, 32, 40, 48 and 52 or premature D/C

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (5):
  - Rush University Medical Center, Chicago, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - Hepatobiliary Associates of New York, Bayside, New York
  - Liver Associates of Texas, Houston, Texas
  - Liver Specialist of Texas, Houston, Texas
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico